CLINICAL TRIAL: NCT06182566
Title: A Pilot Randomized Trial of Hybrid Persistent Atrial Fibrillation Ablation in Heart Failure CONVERGE-HF
Brief Title: Hybrid Persistent Atrial Fibrillation Ablation in Heart Failure
Acronym: CONVERGE-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Department feasibility
Sponsor: The Cleveland Clinic (Other)
Collaborators: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Withdrawn
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Catheter ablation including PVI and posterior wall ablation
  Interventions: Procedure: Catheter ablation
- Intervention (Experimental): Convergent ablation Surgical epicardial ablation/ LAA clip/ ablation of ligament of Marshall Catheter Ablation including PVI and posterior wall ablation
  Interventions: Procedure: Convergent ablation

INTERVENTIONS:
Procedure: Convergent ablation — Staged hybrid ablation with CONVERGENT epicardial ablation with ablation of the ligament of Marshall and left atrial appendage clip, followed in second stage by endocardial catheter ablation including pulmonary vein isolation and posterior wall ablation with roof and inferior posterior lines in addition to targeting and touching up any areas with signals at the posterior wall
  Arms: Intervention
Procedure: Catheter ablation — Pulmonary vein isolation using commercially available catheters; including pulmonary vein isolation and posterior wall ablation with roof and inferior posterior lines in addition to targeting and touching up any areas with signals at the posterior wall
  Arms: Control

SUMMARY:
Pilot, randomized, unblinded, feasibility and proof of concept clinical trial randomizing 50 patients in a 1:1 ratio to hybrid ablation or catheter ablation

DETAILED DESCRIPTION:
To determine if a hybrid convergent ablation procedure with atrial appendage clip is superior to catheter ablation in the management of heart failure patients with persistent and longstanding persistent AF.

Hypothesis: Hybrid convergent ablation procedure with atrial appendage clip is superior to catheter ablation in the management of heart failure patients with persistent and longstanding persistent AF in terms of mortality and worsening heart failure, AF rhythm control and improvement in LVEF, quality of life, and 6-minute walk distance.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

* Be >18 years of age
* Provide signed written Informed Consent
* Persistent or longstanding persistent AF
* Heart failure with LV systolic dysfunction (defined as EF<40%) and prior hospitalization for heart failure in the preceding 12 months (randomization will account for 2 strata >30% vs <30% to ensure balanced enrollment)
* Moderate or severe left atrial enlargement (Left atrial diameter>45 mm and not exceeding 60 mm; or indexed LA volume >40 ml/m2 and not exceeding 110 ml/ m2)
* Ability to complete 6 minute walk test
* Negative pregnancy test for female patients of child bearing potential.
* Be eligible for ablation and anti-arrhythmic drugs

Exclusion Criteria:

Subjects must meet none of the criteria:

* Very severe left atrial enlargement with diameter >60 mm or indexed LA Volume >110 mL/m2
* Stroke or myocardial infarction within the preceding 3 months
* Reversible causes of AF such as pericarditis, thyroid disorders, acute alcohol intoxication, recent major surgical procedures, or trauma
* Presently with Valvular Heart disease requiring surgical intervention
* Presently with coronary artery disease requiring surgical or percutaneous intervention
* Early Post-operative AF (within three months of surgery)
* History of AVN ablation
* Liver Failure
* Renal Failure requiring dialysis
* Social factors that would preclude follow up or make compliance difficult.
* Contraindication to the use of appropriate anticoagulation therapy
* Enrollment in another investigational drug or device study.
* Patients with severe pulmonary disease
* Documented intra-atrial thrombus, tumor, or another structural abnormality which precludes ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Composite of Major Adverse Event Rate after blanking period post procedure | Up to 2 years
  Major Adverse Events consist of death from cardiovascular causes, worsening of heart failure defined as hospitalization, visits for IV diuresis or escalation to advanced heart failure therapies; need for continuation of AADs or redo ablation for recurrent arrhythmias beyond the blanking period.

SECONDARY OUTCOMES:
AF burden | up to 2 years
  Percentage of AF out of the total monitored time
Death from cardiovascular causes | up to 2 years
  Occurrence of death from cardiovascular causes
Worsening of Heart Failure | up to 2 years
  Occurrence of worsening of heart failure defined as: hospitalization, visits for IV diuresis or escalation to advanced heart failure therapies
Need for continuation of Antiarrhythmic drug(s) beyond the blanking period | 3 month post procedure up to 2 years
  Occurrence of worsening of heart failure defined as: hospitalization, visits for IV diuresis or escalation to advanced heart failure therapies
Redo ablation beyond the blanking period | 3 month post procedure up to 2 years
  Occurrence of arrhythmia requiring redo ablation
Total number of cardiovascular hospitalizations | Up to 2 years
  Number of cardiovascular-related hospitalizations
Recurrence of AF lasting more than 30 seconds | Up to 2 years
  Number of occurrence of AF lasting more than 30 seconds
Change in distance walked in 6-minute walk test | up to 2 years
  Change in meters walked in 6-minute walk test compared to baseline
Change in MLHF Quality of Life | up to 2 years
  Based on composite score (0-105). Each item is scored in a 6-point Likert Scale (0 = none to 5 = very much), thus the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life.
  Score is compared to baseline.
Change in EF during trial period | up to 2 years
  EF percentage change compared to baseline
All-cause mortality | up to 2 years
  Occurrence of death from all-cause
Unplanned hospitalization due to cardiovascular reasons | up to 2 years
  Occurrence of unplanned hospitalizations for cardiovascular reasons
Worsening heart failure requiring unplanned hospitalization or escalation to advanced heart failure therapies | up to 2 years
  Occurrence of worsening heart failure requiring unplanned hospitalization or escalation to advanced heart failure therapies requiring: LV mechanical assist devices, transplant, intravenous inotropes
Cerebrovascular accidents | up to 2 years
  Occurrence of cardiovascular accidents

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Hussein, MD, Principal Investigator — The Cleveland Clinic